CLINICAL TRIAL: NCT04082754
Title: A Clinical Study to Test the Safety, Exposure, and Pharmacodynamic Markers of CSL311 in Subjects With Mild-to-moderate Asthma and in Healthy Volunteers
Brief Title: A Clinical Study to Test the Safety, Exposure, and Pharmacodynamic Markers of CSL311 in Patients With Mild-to-moderate Asthma and in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL311_1001; 2019-001135-32 (EudraCT Number)
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- CSL311 Cohort A1 (SAD Dose 1) (Experimental): Human beta common receptor antagonist monoclonal antibody administered intravenously at a Single Ascending Dose (SAD)
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort A2 (SAD Dose 2) (Experimental): Human beta common receptor antagonist monoclonal antibody administered intravenously at a SAD
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort A3 (SAD Dose 3) (Experimental): Human beta common receptor antagonist monoclonal antibody administered intravenously at a SAD
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort A4 (SAD Dose 4) (Experimental): Human beta common receptor antagonist monoclonal antibody administered intravenously at a SAD
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort A5 (SAD Dose 5) (Experimental): Human beta common receptor antagonist monoclonal antibody administered intravenously at a SAD
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort A6 (SAD Dose 6) (Experimental): Human beta common receptor antagonist monoclonal antibody administered intravenously at a SAD
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort A7 (SAD Dose 7) (Experimental): Human beta common receptor antagonist monoclonal antibody administered intravenously at a SAD
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort A8 (SAD Dose 8) (Experimental): Human beta common receptor antagonist monoclonal antibody administered intravenously at a SAD
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort B1 (MAD Dose 1) (Experimental): Human beta common receptor antagonist monoclonal antibody administered intravenously at a MAD
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- Placebo (Placebo Comparator): 0.9% sodium chloride solution administered intravenously
  Interventions: Drug: Placebo
- Placebo (2) (Placebo Comparator): 0.9% sodium chloride solution administered subcutaneously
  Interventions: Drug: Placebo
- CSL311 Cohort C1 (MAD Dose 1) (Experimental): Human beta common receptor antagonist monoclonal antibody administered subcutaneously (SC)
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort C2 (MAD Dose 2) (Experimental): Human beta common receptor antagonist monoclonal antibody administered subcutaneously
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody
- CSL311 Cohort C3 (MAD Dose 3) (Experimental): Human beta common receptor antagonist monoclonal antibody administered subcutaneously
  Interventions: Biological: Human beta common receptor antagonist monoclonal antibody

INTERVENTIONS:
Biological: Human beta common receptor antagonist monoclonal antibody — Human beta common receptor antagonist monoclonal antibody
  Other Names: CSL311
  Arms: CSL311 Cohort A1 (SAD Dose 1); CSL311 Cohort A2 (SAD Dose 2); CSL311 Cohort A3 (SAD Dose 3); CSL311 Cohort A4 (SAD Dose 4); CSL311 Cohort A5 (SAD Dose 5); CSL311 Cohort A6 (SAD Dose 6); CSL311 Cohort A7 (SAD Dose 7); CSL311 Cohort A8 (SAD Dose 8); CSL311 Cohort B1 (MAD Dose 1); CSL311 Cohort C1 (MAD Dose 1); CSL311 Cohort C2 (MAD Dose 2); CSL311 Cohort C3 (MAD Dose 3)
Drug: Placebo — 0.9% sodium chloride, same volume and same duration as CSL311
  Arms: Placebo; Placebo (2)

SUMMARY:
This is a phase 1, first-in-human (FIH), multi-center, randomized, double-blind, placebo-controlled study of CSL311 in patients with mild-to-moderate asthma. The primary objective of this study is to assess the safety and tolerability of single ascending doses (SAD) and multiple ascending doses (MAD) of CSL311.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 65 years of age with diagnosis of mild-to-moderate asthma for Parts A and B. For part C healthy, male or female subjects 18 to 50 years

Exclusion Criteria:

* Oral/parenteral corticosteroids or anti-interleukin-6 therapy within 6 months prior to screening, or any prohibited therapies prior to screening.
* History or presence of clinically significant hypertension or other significant cardiovascular abnormality.
* Any clinically significant abnormality on electrocardiogram at screening.
* Parasitic infestation within 6 months before screening, or travel or intention to travel to a country with a high prevalence of such infections within 1 year before screening or within 85 days after the last dose of CSL311.
* Occurrence of asthma exacerbation and/or upper/lower respiratory tract infection, or any acute infection or disease within the last 6 weeks before screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events (TEAEs) in SC single dose, single ascending doses (SAD) and multiple ascending doses (MAD - SC and IV) | After infusion or injection, up to Day 85 for Cohorts A1 to A7, Day 57 for Cohort A8, Day 114 for Cohort B1 and Day 85 for Cohorts C1 to C3
Percentage of subjects with related TEAEs in SC single dose, SAD and MAD (SC and IV) | After infusion or injection, up to Day 85 for Cohorts A1 to A7, Day 57 for Cohort A8, Day 114 for Cohort B1 and Day 85 for Cohorts C1 to C3
Percentage of subjects with TEAEs by severity in SC single dose, SAD and MAD (SC and IV) | After infusion or injection, up to Day 85 for Cohorts A1 to A7, Day 57 for Cohort A8, Day 114 for Cohort B1 and Day 85 for Cohorts C1 to C3
  Severity of TEAEs defined as mild, moderate, or severe

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of CSL311 in SAD | Up to 85 days after infusion
Time to reach Cmax (tmax) of CSL311 in SAD | Up to 85 days after infusion
Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-last) of CSL311 in SAD | Up to 85 days after infusion
Area under the concentration-time curve from time 0 extrapolated to infinite time (AUC0-inf) of CSL311 in SAD | Up to 85 days after infusion
Half-life (t½) of CSL311 in SAD | Up to 85 days after infusion
Clearance (CL) of CSL311 in SAD | Up to 85 days after infusion
Volume of distribution (Vd) of CSL311 in SAD | Up to 85 days after infusion
Area under the concentration-time curve from time 0 to the last measurable concentration per dose of CSL311 (AUC0-last/dose) in SAD | Up to 85 days after infusion
Cmax/dose of CSL311 in SAD | Up to 85 days after infusion
AUCtau for CSL311 in MAD (SC and IV) after first dose | Up to 15 days after infusion or injection
AUCtau/dose for CSL311 in MAD (SC and IV) after first dose | Up to 15 days after infusion or injection
Cmax of CSL311 in MAD (SC and IV) after first dose | Up to 15 days after infusion or injection
Cmax/dose of CSL311 in MAD (SC and IV) after first dose | Up to 15 days after infusion or injection
  Dose-normalized maximum plasma concentration
tmax of CSL311 in MAD (SC and IV) after first dose | Up to 15 days after infusion or injection
Cmax of CSL311 in MAD (SC and IV) after last dose | Up to 85 days (SC) and 114 days (IV) after infusion or injection
AUCtau for CSL311 in MAD (SC and IV) after last dose | Up to 85 days (SC) and 114 days (IV) after infusion or injection
Cmax/dose of CSL311 in MAD (SC and IV) after last dose | Up to 85 days (SC) and 114 days (IV) after infusion or injection
tmax of CSL311 in MAD (SC and IV) after last dose | Up to 85 days (SC) and 114 days (IV) after infusion or injection
AUCtau/dose for CSL311 in MAD (SC and IV) after last dose | Up to 85 days (SC) and 114 days (IV) after infusion or injection
  Dose-normalized area under the concentration-time curve over a dosing interval
Half-life (t½) of CSL311 in MAD (SC and IV) after last dose | Up to 85 days (SC) and 114 days (IV) after infusion or injection
Clearance (CL) of CSL311 in MAD (IV) after last dose | Up to 114 days after infusion
Apparent Clearance (CL/F) of CSL311 in MAD (SC) after last dose | Up to 85 days after injection
Volume of distribution (Vd) of CSL311 in MAD (IV) after last dose | Up to 114 days after infusion
Apparent volume of distribution during terminal phase (Vz/F) of CSL311 in MAD (SC) after last dose | Up to 85 days after injection
Number of subjects with detectable anti-CSL311 antibodies in SAD and MAD (SC and IV) | After infusion or injection, up to 85 days for SAD, and up to 85 days for MAD (SC) and 114 days for MAD (IV)
Percentage of subjects with TEAEs of Infections and Infestations in SAD and MAD (SC and IV) by treatment (CSL311 or placebo), by causality, and by CSL311 dose level | After infusion or injection, up to 85 days for SAD, and up to 85 days for MAD (SC) and 114 days for MAD (IV)
Percentage of subjects with severe or life-threatening Neutropenia in SAD and MAD (SC and IV) by treatment (CSL311 or placebo), by causality, and by CSL311 dose level | After infusion or injection, up to 85 days for SAD, and up to 85 days for MAD (SC) and 114 days for MAD (IV)
Percentage of subjects with TEAEs of Worsening Asthma in SAD and MAD (SC and IV) by treatment (CSL311 or placebo), by causality, and by CSL311 dose level | After infusion or injection, up to 85 days for SAD, and up to 85 days for MAD (SC) and 114 days for MAD (IV)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (3):
- Germany (2):
  - Paraxel Berlin, Berlin
  - Fraunhofer-Institut für Toxikologie und Experimentelle Medizin ITEM, Hanover
- Medicines Evaluation Unit, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.